CLINICAL TRIAL: NCT02738567
Title: Assessment of Adverse Cardiac Events Using Local Anesthesia With Adrenaline
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0277-15-MMC
Record Dates: First submitted 2016-04-03; First posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Arrythmia
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- local anesthesia with adrenaline: patients undergoing surgery or medical procedure with the use of local anesthesia with adrenaline
  Interventions: Procedure: patients undergoing surgery or medical procedure
- local anesthesia without adrenaline: patients undergoing surgery or medical procedure with the use of local anesthesia without adrenaline
  Interventions: Procedure: patients undergoing surgery or medical procedure

INTERVENTIONS:
Procedure: patients undergoing surgery or medical procedure

SUMMARY:
The use of vasopressor supplement materials to local anesthetics is commonly used in procedures in various fields of dentistry, ENT (ear, nose, and throat), Plastic Surgery, Hand surgery and gastroenterology. Epinephrine is used to constrict small blood vessels, thus reducing bleeding during a medical procedure, reducing the toxicity by reducing systemic absorption of local anesthetic, and prolonging the duration and intensity of neural blockage created by the local anesthetic.

There are descriptions in the literature of cases in which the use of lidocain and adrenaline caused adverse cardiac events such as arrhythmias, edema and increase in blood pressure during ENT and dentistry procedures. As far as we know there has never been a systematic examination of the incidence and severity of arrhythmias during procedures with local anesthesia.

The purpose of the study:

1. To examine the prevalence and types of arrhythmias in patients undergoing a medical procedure performed under local anesthesia
2. Examine whether adding adrenaline to the local anesthetics affects the incidence of arrhythmia Determining the prevalence and types of arrhythmia will help determine the need for monitoring and type of monitoring required during procedures under local anesthesia.

The patients:

500 patients undergoing surgery or a medical procedure in which a local anesthetic is used at Meir Hospital. Patients with a medical history of known cardiac arrhythmia will not be included.

Methods:

Patients will undergo the medical procedure prescribed for them, using local anesthesia with or without adrenaline, at the discretion of the surgeon, in accordance with the usual routine being applied nowadays. The amount and type of anesthesia used will be registered. In addition to the routine monitoring that is currently performed (blood pressure cuff and non-invasive blood oxygen saturation) a continuous ECG monitoring device will be connected prior to the beginning of the surgical procedure, until the patient is discharged from the recovery room. The ECG monitoring results will be analyzed to detect arrhythmia. Side effects being reported by patients (palpitations, dizziness, fainting, CPR {cardiopulmonary resuscitation} ) will be recorded. In cases that an arrhythmia is detected, the type of arrhythmia and the presence of clinical symptoms will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing surgery or a medical procedure in which a local anesthetic is used at Meir Hospital.

Exclusion Criteria:

* Patients with a medical history of known cardiac arrhythmia will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients undergoing surgery or a medical procedure in which a local anesthetic is used at Meir Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
number of participants with arrythmia | day 1

IPD SHARING:
Plan to Share IPD: No